CLINICAL TRIAL: NCT00432705
Title: Modulation of Sensorimotor Measures in Chronically Unstable Ankles
Brief Title: Changes in Unstable Ankles After Balance Training
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Charlotte (Other)
Responsible Party: JoEllen Sefton, UNCCharlotte
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-11-34-CAI-B
Record Dates: First submitted 2007-02-06; First posted 2007-02-08 (Estimated); Last update posted 2009-07-22 (Estimated); Status verified 2009-07

CONDITIONS: Ankle Injury
Keywords: ankle; sensorimotor; reflex; training
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Checking stability of ankle — Flexing and walking
  Other Names: Flexibility study

SUMMARY:
This study is evaluating reflex board training to see if it will help people who frequently roll their ankles. We are investigating several tests that evaluate the ability of the neuromuscular system to control ankle movement. This study is in 2 parts:Part 1 looks at changes after 1 day of reflex training; Part 2 looks at changes after 6 weeks of reflex training. It is thought that the reflex training will improve measures of static and dynamic balance as well as spinal reflex measures.

DETAILED DESCRIPTION:
Research has utilized multiple measures in an effort to detect chronic ankle instability (CAI). Recently, investigations have focused on assessment of sensorimotor function in those who suffer from CAI. These measures have included traditional and functional postural control variables, as well as measures of joint position sense, neuromuscular control and recruitment, and nerve conduction velocity. This study seeks to modulate sensorimotor measures through both short- and long-term reflex training. This information may help to better assess sensorimotor deficits associated with CAI, to focus future research, evaluate rehabilitation protocols and to improve our understanding of this chronic disability.

ELIGIBILITY:
Inclusion Criteria:

* chronically unstable ankles with a history of at least 2 ankle sprains in the past year, M/F 18-30, healthy

Exclusion Criteria:

* ankle sprain within past 6 months, any chronic lower extremity injury or condition, neurological condition, balance-inner ear or vestibular condition, any other condition that would interfere with testing

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2006-09; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
postural control | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: JoEllen M. Sefton, MS, ATC, CMT, Principal Investigator — UNC Charlotte